CLINICAL TRIAL: NCT06700915
Title: A Clinical Trial to Assess the Efficacy and Tolerance of a Berberine-based Nutraceutical Formula to Aid Blood Sugar Regulation and Metabolism
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Ultimate International, Inc. (Industry)
Collaborators: Citruslabs (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 20442
Record Dates: First submitted 2024-11-07; First posted 2024-11-22 (Actual); Last update posted 2024-12-13 (Actual); Status verified 2024-12

CONDITIONS: Metabolism Disorder; Nutraceutical
Keywords: Blood Sugar Regulation; Berberine
MeSH Terms: conditions — Metabolic Diseases

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Diaberine (Experimental): Participants in this arm will receive the Diaberine supplement, which contains Vitamin B12, berberine, magnesium citrate, water-extracted cinnamon bark (Cinnamomum cassia) at a 10:1 ratio, chromium (picolinate), rice flour, dicalcium phosphate, l-leucine, and HPMC (capsule).
  Interventions: Dietary Supplement: Diaberine
- Placebo (Placebo Comparator): Participants in this arm will receive a placebo capsule containing rice flour, dicalcium phosphate, l-leucine, and HPMC (capsule).
  Interventions: Dietary Supplement: Placebo Capsule

INTERVENTIONS:
Dietary Supplement: Diaberine — Participants will take one capsule three times daily, 15 minutes prior to meals, over a 24-week period.
  Arms: Diaberine
Dietary Supplement: Placebo Capsule — Participants will take one capsule three times daily, 15 minutes prior to meals, over a 24-week period.
  Arms: Placebo

SUMMARY:
This randomized, triple-blind, placebo-controlled study will evaluate the efficacy of Diaberine, a berberine-based nutraceutical, in aiding blood sugar regulation and metabolism in 80 participants over 24 weeks.

ELIGIBILITY:
Inclusion Criteria:

* Male or female.
* BMI: 27-35 kg/m2
* HbA1c of 5.7%-6.4% (determined by prescreening blood test)
* Be generally healthy
* Willing to refrain from taking any products, prescription medications, or supplements that target blood sugar regulation or metabolism during the test period.
* Willing to maintain their current diet, sleep schedule, and activity level for the duration of the study.

Exclusion Criteria:

* Diagnosed with Type 2 diabetes mellitus (T2DM) and have been prescribed metformin, insulin, Sulfonylureas, Meglitinides, SGLT2 inhibitors and/or GLP-1 medications including the following prescription medications: Wegovy (semaglutide), Ozempic (semaglutide), Rybelsus (semaglutide), Saxenda (liraglutide), Victoza (liraglutide), Zepbound (bimagrumab), Byetta (exenatide), Bydureon (exenatide ER), Trulicity (dulaglutide), Adlyxin (lixisenatide)
* Current use or past history of use within the last 2 months (8 weeks) of the following prescription medications: Beta-blockers Sectral (Acebutolol), Tenormin (Atenolol), Kerlone, Betoptic (Betaxolol), Zebeta (Bisoprolol), Coreg, Coreg CR (Carvedilol), Trandate, Normodyne (Labetalol), Lopressor, Toprol XL (Metoprolol), Corgard (Nadolol), Bystolic (Nebivolol), Levatol (Penbutolol), Visken (Pindolol), Inderal, Inderal LA, InnoPran XL (Propranolol). Thiazide diuretics Diuril (Chlorothiazide), Microzide (Hydrochlorothiazide), Thalitone, Hygroton (Chlorthalidone), Lozol (Indapamide), Zaroxolyn (Metolazone), Naturetin (Bendroflumethiazide), Enduron (Methyclothiazide). Corticosteroids Deltasone (Prednisone), Orapred, Prelone (Prednisolone), Medrol (Methylprednisolone), Qvar (Beclomethasone), Celestone (Betamethasone), Decadron (Dexamethasone), Cortef (Hydrocortisone), Kenalog (Triamcinolone). Immunosuppressants Tacrolimus (Prograf), Cyclosporine (Neoral), Sirolimus (Rapamune)
* Women who are pregnant, breastfeeding, or trying to conceive.
* Anyone unwilling or unable to follow the study protocol.
* Any pre-existing chronic conditions that would prevent participants from adhering to the protocol, including oncological and psychiatric disorders.
* Is currently undergoing or planning to undergo any significant medical procedures in the next six months
* Has had any major illness in the last three months.
* A history of severe allergic reactions, including but not limited to any of the product's ingredients.
* Heavy drinkers or drug users. A heavy drinker is considered to be a woman who drinks 8 or more alcoholic drinks per week or a man who drinks 15 or more alcoholic drinks per week.
* Impaired hepatic function.
* Individuals taking prescription or over-the-counter medication, or herbal remedies that affect blood sugar regulation or metabolism.
* Currently being treated for an infection with an antibiotic and/or antiviral prescription medication.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80 (Estimated)
Dates: Start 2024-10-03 (Actual); Primary Completion 2025-05-01 (Estimated); Study Completion 2025-05-01 (Estimated)

PRIMARY OUTCOMES:
Blood Sugar Regulation | Baseline, Week 12, and Week 24
  Evaluation of the effect of Diaberine on blood sugar regulation as measured by changes in HbA1c
Metabolism | Baseline, Week 12, and Week 24
  Evaluation of the effect of Diaberine on metabolism, as measured by changes in lipid panel levels.

SECONDARY OUTCOMES:
Quality of Life change | Baseline, Week 4, Week 8, Week 12, Week 16, Week 20, and Week 24; Weight: Baseline and Week 24
  Assessment of participant-reported quality of life via a questionnaire.
Weight Change | Baseline, Week 4, Week 8, Week 12, Week 16, Week 20, and Week 24; Weight: Baseline and Week 24
  Evaluation of changes in participant weight.

CONTACTS AND LOCATIONS:
Locations (1):
- Citruslabs, Santa Monica, California, United States

IPD SHARING:
Plan to Share IPD: No